CLINICAL TRIAL: NCT03014323
Title: Racial Differences in Vagal Control of Glucose Homeostasis, Chronic Study
Acronym: RDVCGH
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No fundings
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 141552-specific aim 2
Record Dates: First submitted 2017-01-03; First posted 2017-01-09 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Insulin Sensitivity; Oxidative Stress
Keywords: insulin sensitivity; African American; obese
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Galantamine then Placebo, WW (Experimental): 4 mg (1 capsule) galantamine twice a day for 4 weeks then placebo (1 capsule) twice a day for 4 weeks in white women (WW)
  Interventions: Drug: Galantamine; Drug: Placebo
- Placebo then Galantamine, WW (Placebo Comparator): Placebo (1 capsule) twice a day for 4 weeks then 4 mg (1 capsule) galantamine twice a day for 4 weeks in white women (WW)
  Interventions: Drug: Galantamine; Drug: Placebo
- Galantamine then Placebo, AAW (Experimental): 4 mg (1 capsule) galantamine twice a day for 4 weeks then placebo (1 capsule) twice a day for 4 weeks in African American Women (AAW)
  Interventions: Drug: Galantamine; Drug: Placebo
- Placebo then Galantamine, AAW (Placebo Comparator): Placebo (1 capsule) twice a day for 4 weeks then 4 mg (1 capsule) galantamine twice a day for 4 weeks African American Women (AAW)
  Interventions: Drug: Galantamine; Drug: Placebo

INTERVENTIONS:
Drug: Galantamine — Galantamine 4 mg twice a day for 4 weeks
  Other Names: Razadyne
Drug: Placebo — Placebo 1 capsule twice a day for 4 weeks
  Other Names: Razadyne

SUMMARY:
Investigators will test the hypothesis that chronic restoration of vagal nerve activity with a central acetylcholinesterase inhibitor improves insulin sensitivity and reduces adipose tissue oxidation in obese African American Women compared to white women.

DETAILED DESCRIPTION:
Investigators will test the hypothesis that chronic restoration of parasympathetic nervous system (PNS) activity with a central acetylcholinesterase inhibitor improves insulin sensitivity and reduces adipose tissue oxidation in obese African American women (AAW) compared to white women (WW). A cross-over study will be performed in matched cohorts of AAW and white women subjected to chronic central acetylcholinesterase inhibition with galantamine versus placebo, given orally over a 4-week period. Insulin sensitivity will be measured using the gold standard hyperinsulinemic-euglycemic clamp. Adipose tissue will be obtained through subcutaneous fat biopsies where F2-isoprostanes will be quantified.

ELIGIBILITY:
Inclusion Criteria

* Female
* African American or white (race will be self-defined, but only subjects who report both parents of the same race will be included)
* 18-60 years old
* BMI 30-45 Kg/m2
* Not pregnant or breastfeeding

Exclusion Criteria

* Pregnant or breastfeeding
* Diabetes diagnosis (defined by the American Diabetes Association (ADA) criteria)38
* Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy.
* Arrhythmia (first-, second-, and third-degree AV block)
* Significant weight change >5% in the past 3 months
* Impaired hepatic function (AST and/or ALT >1.5X upper limit of normal range)
* Impaired renal function (eGFR <60ml/min)
* Users of strong inhibitors of CYP3A4 or CYP2D6
* Users of other acetylcholinesterase inhibitors such as pyridostigmine or bethanechol
* History of alcohol or drug abuse
* Mental conditions rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Steroid use within 6 weeks prior to study entry
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Discretion of the investigator

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity | 4 weeks
  insulin sensitivity will be measured with hyperinsulinemic euglycemic clamps

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya A Shibao, MD, Principal Investigator — Vanderbilt University Medical Center, Clinical Pharmacology
Locations (1):
- Cyndya Shibao, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No sharing